CLINICAL TRIAL: NCT04294017
Title: The Soluble VCAM-1 / Soluble ICAM-1 Ratio as a Non-invasive Biomarker for Diagnosing Endometriosis - a Prospective Multicenter Validation Study
Brief Title: CellAdhesionMolecule EndometriosisRatio - CAMERA
Acronym: CAMERA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich Husslein (Other)
Collaborators: Medical-Scientific Fund of the Mayor of the Federal Capital Vienna (Unknown)
Responsible Party: Sponsor-Investigator, Heinrich Husslein, Assoc.Prof.Priv.Doz Dr.med.univ. , PLL.M., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1496/2017
Record Dates: First submitted 2020-01-24; First posted 2020-03-03 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Endometriosis (Diagnosis); Identification of Biomarkers in Serum
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Up to 4 ml of serum per participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: participants undergoing a diagnostic laparoscopy and have a histologically confirmed Endometriosis
- controls: participants undergoing a diagnostic laparoscopy where no evidence of Endometriosis could be found

SUMMARY:
Background: Endometriosis, which is characterized by the growth of endometrial stroma and glands outside of the uterine cavity, is estimated to occur in 6-10% of women of reproductive age. Clinical presentation of endometriosis can vary widely, often significantly reducing quality of life, and the mean interval between the onset of symptoms and obtaining a definitive diagnosis is approximately 10 years. Currently, laparoscopy is the gold standard for diagnosing endometriosis; however, this procedure is invasive, carries surgery-related risks, and contributes to diagnostic delay. Therefore, the field has an urgent need for an efficient, sensitive, non-invasive tool for diagnosing endometriosis.

Recently, it was shown that sVCAM-1/sICAM-1 ratio is a promising serum biomarker, which may lead to the development of a new, efficient, sensitive, non-invasive tool for diagnosing endometriosis, thereby potentially avoiding surgical interventions.

Primary aim: To determine whether the serum sVCAM-1/sICAM-1 ratio can be used todiagnose endometriosis.

Study design: Prospective multicenter validation study

ELIGIBILITY:
Inclusion Criteria:

* unfulfilled desire for children
* chronic pelvic pain
* suspicion of endometriosis
* cysts
* myomas

Exclusion Criteria:

* acute infections
* malign diseases
* drug abuse
* pregnancy
* infectious diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women in reproductive age undergoing a diagnostic laparoscopy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
sICAM and sVCAM in serum | up to 1 week
  levels of these two soluble adhesion factors in serum of patients and controls

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria